CLINICAL TRIAL: NCT03199261
Title: The Pharmacokinetic Comparison and Bioequivalence Evaluation of Two 10-µg Recombinant Exendin-4 Formulations in Chinese Healthy Male Subjects
Brief Title: A Study of Pharmacokinetic Comparison of Two Recombinant Exendin-4 Formulations in Chinese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SN-YQ-2016018
Record Dates: First submitted 2017-01-17; First posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2016-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rE-4 Injection (Experimental): 10µg, rE-4 Injection, 30 minutes prior to the start time of a standard breakfast.
  Interventions: Drug: rE-4 Injection
- rE-4 Freeze-dried Powder (Active Comparator): 10µg, rE-4 Freeze-dried Powder, 30 minutes prior to the start time of a standard breakfast.
  Interventions: Drug: rE-4 Freeze-dried Powder

INTERVENTIONS:
Drug: rE-4 Injection — During the study session, healthy subjects will be receive a subcutaneous single dose of rE-4 Injection 10µg administered 30 minutes prior to the start time of a standard breakfast.
  Other Names: Recombinant Exendin-4 Injection
  Arms: rE-4 Injection
Drug: rE-4 Freeze-dried Powder — During the study session, healthy subjects will be receive a subcutaneous single dose of rE-4 Freeze-dried Powder 10µg administered 30 minutes prior to the start time of a standard breakfast.
  Other Names: Recombinant Exendin-4 Freeze-dried Powder
  Arms: rE-4 Freeze-dried Powder

SUMMARY:
Evaluation of the pharmacokinetics and safety rE-4 Injection versus rE-4 Freeze-dried Powder in healthy subjects.

DETAILED DESCRIPTION:
The study design is an Open-Label Randomized, Single-Dose, 2-way Crossover Bioequivalence Study with a washout period of 7 days. During each session, the subjects will receive a subcutaneous single dose of rE-4 (rE-4 Injection 10µg or rE-4 Freeze-dried Powder 10µg) administered 30min prior to the start time of a standard breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adult volunteers of 18-45 years old, who can be inserted needle.
* Body mass index (BMI) of 19 to 26 kg/m2, inclusive BMI = weight (kg)/[height(m)]2，During Screening period body weight≥50 kg.
* Subjects are fully informed and voluntarily consent to participate in this study.

Exclusion Criteria:

* A positive result in hepatitis B surface antigen (HBsAg), hepatitis B e antigen (HBeAg), anti-hepatitis C virus (HCV) antibodies, a syphilis test, or an human immunodeficiency virus (HIV) test.
* History or presence of neurological, cardiovascular, renal, hepatic, pancreatic,gastrointestinal, pulmonary, metabolic, or musculoskeletal diseases.
* History or presence neurological disorder disease.
* Abnormal laboratory profiles, routine inspection, vitl signs and ECGs results with clinical significance.
* Participation in a clinical drug study 30 days prior to present study.
* FPG≥6.1mmol/L or <3.9mmol/L.
* SBP<90mmHg or >140mmHg; DBP>90mmHg.
* Use of any other drugs,vitamine and mineral substance.
* Blood donation more than 200 mL blood within 3 months prior to the study.
* Smoker (>5 cigarettes/day) or alcoholist (355 ml alcohol/day).
* History or Family history of hypoglycemia.
* History of allergy or hypersensitivity.
* Subjects planning to give birth or donate sperm during the study or within 3 months after the study.
* Other unfavorable factors diagnosed by investigators.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12-23; Primary Completion 2017-01-21 (Actual); Study Completion 2017-01-21 (Actual)

PRIMARY OUTCOMES:
Bioequivalency between the 2 formulations of rE-4 | before injection and 0.25,0.5,0.75,1.0,1.5，2.0,3.0,4.0,6.0,8.0hour post-injection
  Area under curve

CONTACTS AND LOCATIONS:
Overall Officials: Hengyan Qu, Ph.D, Principal Investigator — The Affiliated Hospital Military Medical Sciences
Locations (1):
- The Affiliated Hospital Military Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No